CLINICAL TRIAL: NCT00100061
Title: Dose Response to Cranberry of Women With Recurrent UTIs
Brief Title: Effects of Cranberry-Containing Products in Women With Recurrent Urinary Tract Infections (UTIs)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Collaborators: Office of Dietary Supplements (ODS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R01AT002090-01 (NIH)
Record Dates: First submitted 2004-12-22; First posted 2004-12-23 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Urinary Tract Infection
Keywords: Cranberry; Vaccinium macrocarpon
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cranberry Juice (Active Comparator): Cranberry Juice provided by Ocean Spray
  Interventions: Drug: Cranberry juice; Dietary Supplement: Cranberry Juice
- Placebo cranberry juice (Placebo Comparator): Taken orally
  Interventions: Dietary Supplement: Placebo cranberry juice

INTERVENTIONS:
Drug: Cranberry juice — liquid juice taken daily
  Arms: Cranberry Juice
Dietary Supplement: Cranberry Juice — Taken orally
  Arms: Cranberry Juice
Dietary Supplement: Placebo cranberry juice — Placebo comparitor
  Arms: Placebo cranberry juice

SUMMARY:
The purpose of this study is to determine the role of cranberry-containing products in preventing urinary tract infections (UTIs).

DETAILED DESCRIPTION:
Although cranberry-containing products are commonly taken to prevent UTIs and other urinary symptoms, an optimally effective dose has not been established, and the chemicals responsible for the UTI-preventing properties in cranberry-containing products have yet to be determined. This study will determine the minimum dose of cranberry-containing product necessary to prevent UTIs, the effectiveness of cranberry-containing products in fighting different strains of E. coli, and the long-term effects of cranberry-containing product consumption. This study will also determine whether plant pigments called proanthocyanidins influence the UTI-preventing properties of cranberry-containing products.

This study will last 2 years. Participants will be randomly assigned to receive varying doses of either cranberry-containing products or placebo for 1 year. Some participants will receive cranberry or placebo supplement tablets; others will receive cranberry juice or a placebo beverage. Clinic visits will occur every 2 months; urine collection will occur at each visit. Some participants will be asked to collect 24-hour urine samples every 8 weeks and provide urine samples on Days 1, 3, 5 and 7.

Laboratory tests will be used to assess participants during the study. A 3-day course of antibiotics will be provided to participants developing a UTI during the course of the study. Telephone interview follow-up at 6 and 12 months after the study will determine whether cranberry-containing product use has continued and whether UTIs have recurred.

ELIGIBILITY:
Inclusion Criteria:

* At least two UTIs in the year prior to study entry
* Willing to use acceptable methods of contraception
* Willing to refrain from consuming other forms of cranberry supplementation

Exclusion Criteria:

* Current UTI
* Allergy to cranberry-containing products
* Active urinary stone disease
* Insulin-dependent diabetes
* Immunosuppressive disease
* Current corticosteroid use
* Intermittent or indwelling catheterization
* Pregnancy

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2007-05; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Minimum dose of cranberry-containing product necessary to achieve a 30% prophylaxis of UTIs in women with recurrent UTIs | end of study
  recurrence of UTI
Whether the degree of UTI prophylaxis is related to the dose of cranberry-containing product (dose response curve) | end of study
  comparison of UTI occurrence
Whether proanthocyanidin concentration in the urine correlates with UTI prophylaxis | end of study
  recurrence of UTI and lab results

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Stothers, MD, Principal Investigator — Bladder Care Centre, University of British Columbia
Locations (1):
- Bladder Care Centre, University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Williams G, Stothart CI, Hahn D, Stephens JH, Craig JC, Hodson EM. Cranberries for preventing urinary tract infections. Cochrane Database Syst Rev. 2023 Nov 10;11(11):CD001321. doi: 10.1002/14651858.CD001321.pub7. PMID 37947276
- [Derived] Williams G, Hahn D, Stephens JH, Craig JC, Hodson EM. Cranberries for preventing urinary tract infections. Cochrane Database Syst Rev. 2023 Apr 17;4(4):CD001321. doi: 10.1002/14651858.CD001321.pub6. PMID 37068952